CLINICAL TRIAL: NCT02551614
Title: Measurement of Neutrophil Retention in the Lung in Vivo, Using Autologous Labelled Neutrophils, in Healthy Subjects Following Lipopolysaccharide or Saline Challenge and Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Neutrophil Imaging in Healthy Subjects Following Lipopolysaccharide or Saline Challenge and in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201463
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: lipopolysaccharide; COPD; neutrophil
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: healthy subjects (Experimental): Subjects will undergo inhaled challenge, either with lipopolysaccharide or saline in a 2:1 ratio, prior to imaging assessments. Assessments will be performed during one study day on an outpatient basis.
  Interventions: Procedure: Lipopolysaccharide challenge; Procedure: Saline challenge; Procedure: Labelled neutrophils and Imaging assessment
- Group 2: COPD patients (Experimental): Subjects will undergo imaging assessments during one study day on an outpatient basis. Approximately 10 of these COPD patients will repeat this study day 7-10 days after completion of the first study day to assess the reproducibility of the technique.
  Interventions: Procedure: Labelled neutrophils and Imaging assessment

INTERVENTIONS:
Procedure: Lipopolysaccharide challenge — Lipopolysaccharide solution inhaled using a dosimeter.
  Arms: Group 1: healthy subjects
Procedure: Saline challenge — 0.9% sodium chloride solution inhaled using dosimeter.
  Arms: Group 1: healthy subjects
Procedure: Labelled neutrophils and Imaging assessment — Injection of labelled neutrophils and imaging assessments

SUMMARY:
This is an exploratory study to further develop an imaging platform for the assessment of whole lung neutrophil retention. The primary objective of the study is to quantify and compare neutrophil retention in the lungs of lipopolysaccharide-challenged healthy subjects, saline-challenged healthy subjects and subjects with stable COPD. There will be two treatment groups, one with healthy subjects and the other with subjects with stable COPD. The total duration of this study for healthy subjects will be approximately 1 week, in addition to the screening window of 28 days. The total duration of this study for subjects with COPD will be approximately 1 week for those that complete Visit 1 only, and approximately 2 weeks for those subjects with COPD that return to the unit for Visit 2 7-10 days later, in addition to the screening window of 28 days.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Healthy subjects

* Between 45 and 75 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring:

A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

A subject with well-controlled hypertension, non-insulin dependent diabetes or other well controlled medical conditions may be included if the investigator, in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects must be stable on their current treatment for at least one month prior to first imaging visit.

* Current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of less than 5 pack years.

Pack years = (cigarettes per day smoked/20) x number of years smoked)

* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19-30 kg/meter (m)^2 (inclusive).
* Males.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative human chorionic gonadotrophin (hCG) test), not lactating, and of non reproductive potential defined as:

Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Group 2: COPD patients

* Between 45 and 75 years of age inclusive, at the time of signing the informed consent.
* Stable stage 2-3 COPD patients, in accordance with the definition in the GOLD guidelines, 2014 and with forced expiratory volume in one second (FEV1) >=40% predicted. Stable is defined as: No COPD exacerbations in the 3 months prior to first imaging visit. Subjects who are stable on their current treatment for at least one month prior to first imaging visit.
* Body weight >=45 kg and BMI within the range 18-32 kg/m^2 (inclusive).
* Males
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative hCG test), not lactating, and of non reproductive potential defined as:

Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with FSH and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on HRT and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

Group 1: healthy subjects

* Alanine aminotranseferase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QT corrected by Frederica's formula (QTcF) >450 millisecond (msec).
* History of acute respiratory illnesses within 4 weeks prior to screening.
* Asthma or history of asthma (including seasonal asthma).
* Oxygen saturation below 94% on room air.
* Spirometry FEV1 <=80% of predicted or FEV1/FVC ratio <=70% at screening.
* Ongoing treatment with statins that will be continued during the study or within two weeks of the first imaging visit.
* History of regular alcohol consumption within 6 months of the study defined as: For United Kingdom sites: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (equivalent to 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to the study challenge agent, radiochemicals, or components thereof, or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained.
* A positive pre-study smoking/drug/alcohol screen.
* A positive test for human immunodeficiency virus antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first imaging visit in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first imaging visit.
* Previous exposure to ionising radiation above background (e.g. through work or research studies) that, combined with the estimated exposure dose to be given in this study, results in exposure over 10Milisievert (mSv) in a three year period. Clinical (therapeutic or diagnostic) exposures or those that involve patient benefit will not be included in this calculation.

Group 2: COPD patients

* ALT and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF > 450 msec or QTcF > 480 msec in subjects with Bundle Branch Block
* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, pulmonary fibrosis, asthma or any other respiratory condition that might, in the opinion of the Investigator, compromise the safety of the or affect the interpretation of the results.
* Any other concurrent inflammatory condition.
* Anemia until adequately treated.
* Ongoing treatment with monoclonal antibodies or treatment with monoclonal antibodies in the 12 months prior to the first imaging visit.
* Ongoing treatment with systemic corticosteroids or systemic corticosteroids within 6 weeks prior to first imaging visit.
* History of regular alcohol consumption within 6 months of the study defined as: For United Kingdom sites: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (equivalent to 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to the radiochemicals, or components thereof, or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of HBsAg, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA PCR test is obtained.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the imaging visit in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first imaging visit.
* Previous exposure to ionising radiation above background through research studies or work that, combined with the estimated exposure dose to be given in this study, results in exposure over 10mSv in a three year period. Clinical (therapeutic or diagnostic) exposures or those that involve patient benefit will not be included in this calculation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Uptake of labelled neutrophils in the lung as assessed by single-photon emission tomography (SPECT). | Blood samples will be collected and imaging assessments will be completed after injection of labelled neutrophils at visit 1 (one day) for healthy subjects and visit 1 and 2 (upto two days, 10 days apart) for subjects with COPD.
  Uptake of labelled neutrophils in lungs will be assessed to quantify neutrophil retention in the lungs of healthy subjects, lipopolysaccharide -challenged healthy subjects and subjects with stable COPD.
Comparison of neutrophil lung retention between saline-challenged and lipopolysaccharide -challenged healthy subjects. | Blood samples will be collected and imaging assessments will be completed after injection of labelled neutrophils at visit 1 (one day as an outpatient visit).
Comparison of neutrophil lung retention between COPD patients and saline-challenged healthy subjects. | Blood samples will be collected and imaging assessments will be completed after injection of labelled neutrophils at visit 1 (one day) for healthy subjects and visit 1 and 2 (upto two days, 10 days apart) for subjects with COPD.
Comparison of neutrophil lung retention between COPD patients and lipopolysaccharide -challenged healthy subjects. | Blood samples will be collected and imaging assessments will be completed after injection of labelled neutrophils at visit 1 (one day) for healthy subjects and visit 1 and 2 (upto two days, 10 days apart) for subjects with COPD.

SECONDARY OUTCOMES:
Uptake of neutrophils in the lung as assessed by SPECT analysis in stable COPD patients scanned on a second visit, 7-10 days after the first visit. | Blood samples will be collected and imaging assessments will be completed after injection of labelled neutrophils at visit 2 (upto two days as outpatient visits, upto 10 days apart) for subjects with COPD.
  Uptake of labelled neutrophils in lungs will be assessed to investigate the reproducibility of the uptake of labelled neutrophils in subjects with stable COPD.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- [Derived] Tregay N, Begg M, Cahn A, Farahi N, Povey K, Madhavan S, Simmonds R, Gillett D, Solanki C, Wong A, Maison J, Lennon M, Bradley G, Jarvis E, de Groot M, Wilson F, Babar J, Peters AM, Hessel EM, Chilvers ER. Use of autologous 99mTechnetium-labelled neutrophils to quantify lung neutrophil clearance in COPD. Thorax. 2019 Jul;74(7):659-666. doi: 10.1136/thoraxjnl-2018-212509. Epub 2019 Jan 23. PMID 30674586
- See also: Results for study 201463 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201463?search=study&search_terms=201463#rs